CLINICAL TRIAL: NCT05711511
Title: Radiographic Comparison of Obturation Performed by Conventional Method and Obtura II.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, sheejia asif, Principal investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOD/ERB/2022/15
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Tooth Disease
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coventional obturation technique (Experimental): In conventional method, paper point will be used to coat the walls of the canal with sealer, Standardized Protaper F-3 master gutta-percha cone will slid to the working length and ISO No.25 finger spreader was applied under vertical loading.The first accessory cone will slid promptly to proper length with a light coating of sealer. Compaction and accessory cone insertion will be continued;each spreader insertion will be seen to be slightly less deep than former, as mirrored by shorter and shorter accessory cone insertion. Condensation continued until the spreader reached 2-3 mm into the canal. Heat will be applied with to the root filling at or below canal orifice level, and the filling will then compacted apically with the help of a cold plugger.
  Interventions: Procedure: conventional obturation technique; Device: Obtura II
- Obtura II (Active Comparator): The Obtura II system will be prepared ,sealer will be applied to canal wall . A 23G needle is selected and a stopper will place at 4-6 mm of the WL. The control unit of Obtura II will be on, and the display showed the required temperature of 185°C. The gun will be loaded with a fresh pellet of gutta- percha and plunger will be pushed forward.The needle will be then positioned in the canal so that it reached 3 to 5 mm of the apical preparation. 3-4 mm of the gutta-percha was passively injected without any apical pressure and will be compacted gently with a #11 endodontic plugger. Thus, the apical plug will be created in this manner. A segmental technique will be used in which 3 to 4 mm of gutta-percha will be sequentially injected and compacted. Increments will be added until gutta-percha reached top orifice level, and then compaction will be done with a cold plugger. Excess gutta-percha was severed at or below the orifice level.
  Interventions: Procedure: conventional obturation technique; Device: Obtura II

INTERVENTIONS:
Procedure: conventional obturation technique — cold lateral condensation ,this technique involves placing a single cone of gutta-percha (GP) with sealer in the prepared root canal and adding secondary GP cones that are compacted together with the use of a spreader. The cones stay together due to frictional grip and the presence of a sealer
Device: Obtura II — is a popular warm gutta-percha technique that uses a "gun" to warm and inject the gutta-percha filling into the root canal.Obtura 2 system: The gutta-percha is heated from temperature range of 160C to 200C which is then injected through the needle

SUMMARY:
Root canal therapy plays an importanmt role in dental health care.An importanat parameter necessary to achieve a proper endodontic treatment is quality of root canal filling.This study compare the radiographic quality of obturation with cold lateral condensation and thermoplasticiszed gutta percha technique and obtura II system.

DETAILED DESCRIPTION:
The aim of this study is to assess and compare the radiogrphic quality of obturation with thermoplasticized injectable gutta percha technique obtura II system and cold lateral compaction technique in permanent teeth.For this study selected patients will be divided into two groups in a manner that the odd numbers will be alotted to Group A and Group B .Local anesthesia at 2% lidocaineHCl with 1:100000 epinephrine as buccal infiltration in upper teeth and inferior alveolar nerve block in the lower teeth. Access cavity preparation will be done. Canals will be located and negotiated with a DG-16 endodontic explorer . Initial filing will be done from Number 8 to 10 K- files (ISO standardized 0.02 taper) under 5.25% sodium hypochlorite) irrigation and Ethylenediamine Tetra-Acetic Acid as chelating agents.. Working Length will be confirmed with Electronic Apex Locator , and then with working length radiograph will be taken. Rotary preparation will be done with Protaper using S1, S2, F1, F2, F3 files. Master gutta-percha radiograph will be taken at the commencement of the first visit with Protaper F3 gutta-percha point placed in the canals. Intervention will be provided to both groups by the principal investigator. On the second visit, both the canals will be dried with F-3 paper points.Root canal fillings will be then performed using cold lateral condensation in Group A, and thermoplasticized injected gutta-percha in Group B.

Postoperative periapical radiographs will be obtained immediately after the obturation. These radiographs will be examined under illumination in a darkened room at ×2 magnification to assess for voids and termination of obturation. Our study will be based on the radiographic assessment of the buccolingual view of the canals, as it will be the only possible view to visualize on the radiograph in a clinical setting for assessing the quality of endodontic treatment.

Root canal fillings will be assessed

* Presence or absence of voids.
* Acceptable/flush: Root canal filling is within the root canal system and within 2 mm of radiographic apex.
* Under-filled: Root canal filling is >2 mm short of radiographic apex.
* Over-filled: Root canal filling is extruded beyond the radiographic apex

ELIGIBILITY:
Inclusion Criteria:

* Single rooted teeth in which endodontic treatment was clinically indicated.
* Single rooted teeeth in which root canal treatment was recommended for elective reasons.

Exclusion Criteria:

* • Teeth with severely curved roots.

  * Sclerosed canals on periapical radiographs.
  * Periodontally compromised teeth.
  * Endodontic retreatment cases.
  * Teeth with apical resorption.
  * Teeth not salvageable by conventional root canal treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-08-27 (Actual); Primary Completion 2023-02-27 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
optimum extension,overextension ,under extension of obturating material | immediately after the procedure
  radiographically observing the extension of obturating material

SECONDARY OUTCOMES:
Density | immediately after the procedure
  radiographically observing the voids in obturation
adaptation of Gutta percha | immediately after procedure
  radiographically observing the gap between gp and canal wall

CONTACTS AND LOCATIONS:
Overall Officials: sheejia asif, Bds, Principal Investigator — Pims
Locations (1):
- Pims ,school of dentistry, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No